CLINICAL TRIAL: NCT01240486
Title: IMPAACT P1073: Study Of Immune Reconstitution Inflammatory Syndrome (IRIS) For International Sites Initiating Highly Active Antiretroviral Therapy (HAART) In Infants And Children < 72 Months Of Age
Brief Title: IMPAACT P1073: Study of IRIS for Infants and Children Initiating HAART at Int'l Sites
Status: Completed | Type: Observational
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: IMPAACT P1073; U01AI068632 (NIH)
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: IRIS; HIV
Keywords: IRIS; HIV; Immune; Reconstitution; Inflammatory; Syndrome
MeSH Terms: conditions — Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Your child is able to participate in this study, if your child's doctor is planning to start your child on HAART (which is a combination of at least 3 anti HIV drugs). When your child is treated with HAART, the way your child's body is able to fight infection may change. The immune system is the body's defense against infection. Your child's immune system may respond in a stronger way to some types of infections that your child may already have. This immune response may cause your child to become sick and the condition is then called "immune reconstitution inflammatory syndrome" or IRIS.

DETAILED DESCRIPTION:
IMPAACT P1073 is a prospective clinical, observational and pathogenesis study of HIV-infected infants and children who are ART-naïve and will be initiating a HAART regimen at an IMPAACT study site. Where possible, infants and children co-enrolled in IMPAACT studies will be given preference for enrollment in P1073.

The plan is to enroll subjects in P1073 at a timepoint ≤ 1 week prior to starting HAART. For DMC purposes, this is Step 1 for P1073, and subjects are designated as a Non-case, according to the Study Flow Chart

ELIGIBILITY:
Inclusion Criteria

* Past or current documentation of a confirmed diagnosis of HIV-1 infection. Documentation of HIV-1 infection is defined as positive results from two samples collected at different time points. All samples tested must be whole blood, serum, or plasma.

  * Sample #1 may be tested by non-study public or PEPFAR programs. However, both the result and the assay date must be recorded in subject's chart. Source documentation (patient's medical record/chart, Ministry of Health (MOH) registers, laboratory results, etc.) must be available if requested.
  * Sample #2 must be performed in a CAP/CLIA-approved laboratory (for US sites) or in a laboratory that operates according to GCLP guidelines and participates in an appropriate external quality assurance program (for international sites).
  * For P1073, the subject may be enrolled before the result of Sample #2 is available. However, the subject will be taken off study should the 2nd result be negative.

    1. Acceptable tests when subjects are ≤ 18 months of age

       1. Sample #1 may be tested using any of the following: One HIV DNA PCR; One quantitative HIV RNA PCR (>5,000 copies/mL); One qualitative HIV RNA PCR; One total HIV nucleic acid test

          **If Sample #1 is positive, collect and test Sample #2.
       2. Sample #2 may be tested using any of the assays listed above for Sample #1.
    2. Acceptable tests when subjects are > 18 months of age

       1. Sample #1 may be tested using any of the following: Two rapid antibody tests from different manufacturers or based on different principles and epitopes; One EIA OR Western Blot OR immunofluorescence OR chemiluminescence; One HIV DNA PCR; One quantitative HIV RNA PCR (>5,000 copies/mL; One qualitative HIV RNA PCR; One HIV culture (prior to August 2009); One total HIV nucleic acid test

          **If Sample #1 is positive, then collect and test Sample #2.
       2. Sample #2 may be tested using any of the following: One EIA confirmed by Western Blot OR immunofluorescence OR chemiluminescence; One HIV DNA PCR; One quantitative HIV RNA PCR (>5,000 copies/mL); One qualitative HIV RNA PCR; One HIV culture (prior to August 2009;)One total HIV nucleic acid test

          * Rapid antibody tests are not allowed for sample #2
* Age: range is ≥ 4 weeks to < 72 months of age at time of HAART initiation.

  *All infants and children ≥ 4 weeks to < 72 months of age, who are about to initiate HAART according to National or WHO criteria, are eligible.
* HIV-infected infants and children who meet the ART guidelines of local programs or an IMPAACT or other protocol and who can be enrolled ≤ 1 week prior to starting HAART.
* No known active untreated opportunistic infection.
* Infants ≤ 12 months of age should have received BCG immunization and the date of BCG vaccine has to be known.
* Legal guardian able and willing to provide signed informed consent for participating in the IRIS study.

Exclusion Criteria

-Any clinically significant diseases (other than HIV infection) e.g. malignancy, auto-immune or inflammatory diseases requiring long-term immunosuppressive therapy, or clinically significant findings during the screening medical history or physical examination that, in the investigator's opinion, would compromise the outcome of this study. Please contact the team at actg.teamp1073@fstrf.org.

Ages: 4 Weeks to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a prospective, clinical observational and pathogenesis study of HIV-infected infants and children stratified into 2 age groups: ≥ 4 weeks to ≤ 12 months of age; and > 12 to < 72 months of age who will enroll into P1073 at a timepoint ≤ 1 week prior to initiating HAART
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2010-11; Primary Completion 2013-02 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Proportion of study subjects having BCG-related IRIS within 48 weeks of initiating HAART. | within 48 weeks of iniating HAART
Proportion of study subjects having unmasking and paradoxical TB-related IRIS within 48 weeks of initiating HAART. | Within 48 weeks of initiating HAART
Nadir CD4 T-cell count and percentage and plasma viral load pre-HAART initiation, and two weeks post-HAART and CD4 T-cell count and percentage and plasma viral load at the presumptive BCG or TB-IRIS event, for CASES and the matching controls. | At Study Entry, 2 weeks post-HAART and within 48 weeks of initiating HAART
CD4 T-cell count and percentage and plasma viral load, 48 weeks post-HAART initiation for CASES and the matching controls. | 48 weeks post-HAART
Frequency of all IRIS-like events and proportion attributed to BCG or TB. | within 48 weeks of initiating HAART

CONTACTS AND LOCATIONS:
Overall Officials: Mark Cotton, MD, Study Chair — IMPAACT/Stellenbosch University
Locations (7):
- BJ Medical College CRS (31441), Pune, Maharashtra, India
- South Africa (3):
  - Durban Pediatric HIV CRS (20201), Durban, KwaZulu-Natal
  - University of Stellenbosch, Tygerberg Hospital (8950), Cape Town
  - Soweto IMPAACT CRS (8052), Johannesburg
- Kilimanjaro Christian Medical CRS (12901), IDC Research Offices, Moshi, Tanzania
- Makerere University - JHU Research Collaboration (30293), Kampala, Uganda
- UZ-Parirenyatwa CRS (30313), Harare, Zimbabwe